CLINICAL TRIAL: NCT02433288
Title: A Randomized, Two-arm, Open, 24-week Study to Evaluate the Effect of a Smart Phone-based Patient Support Tool on Duration of Treatment in Patients Prescribed Rosuvastatin in China
Brief Title: Rosuvastatin Adherence App Study in China
Acronym: eHELP China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D3560C00088
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-08

CONDITIONS: Dyslipidemia; Hyperlipidemia
Keywords: smart phone-based; rosuvastatin; duration of treatment; Treatment adherence
MeSH Terms: conditions — Dyslipidemias; Hyperlipidemias; Treatment Adherence and Compliance | interventions — Exercise; Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active app (Other): The smart phone application used on the patients' smart phones will contain both the patient support tool and the questions for the clinical evaluation in the form of the Rosuvastatin Adherence questionnaire (RAQ), Beliefs about Medicine Questionnaire - General (BMQ-G), (Horne, 1999) and a Lifestyle questionnaire (LSQ) on disease understanding, lifestyle and treatment awareness. Patients in the Active group will also receive feedback on their daily rosuvastatin treatment as entered in the patient support tool.
  Interventions: Other: Smart phone based patient support tool
- Control app (Other): a smart phone application will be used to prompt patients with the questions for the clinical evaluation (RAQ, BMQ-G and LSQ).
  Interventions: Other: Control application: only for data collection

INTERVENTIONS:
Other: Smart phone based patient support tool — The smart phone application used on the patients' smart phones will contain both the patient support tool and the questions for the clinical evaluation in the form of the Rosuvastatin Adherence questionnaire (RAQ), Beliefs about Medicine Questionnaire - General (BMQ-G), (Horne, 1999) and a Lifestyle questionnaire (LSQ) on disease understanding, lifestyle and treatment awareness. Patients in the Active group will also receive feedback on their daily rosuvastatin treatment as entered in the patient support tool.
  Other Names: Active
  Arms: Active app
Other: Control application: only for data collection — the patients will have no access to the smart phone-based patient support tool. However, a smart phone application will be used to prompt patients with the questions for the clinical evaluation (RAQ, BMQ-G and LSQ).
  Other Names: Control
  Arms: Control app

SUMMARY:
This is a randomized, two-arm, open label, Phase IV clinical trial to evaluate if the provision of a smart phone-based patient support tool prolongs the patient's rosuvastatin treatment duration.

DETAILED DESCRIPTION:
This is a randomised, two-arm, open, Phase IV clinical trial to evaluate if the provision of a smart phone-based patient support tool prolongs the patient's rosuvastatin treatment duration.

Patients diagnosed with dyslipidemia or hyperlipidemia at high risk and are treated with rosuvastatin will be offered participation in the study. Patients who accept and sign the Informed Consent will be randomised into one of two study groups:

* Active group: In this group, patients will have access to the smart phone-based patient support tool. The smart phone application used on the patients' smart phones will contain both the patient support tool and the questions for the clinical evaluation in the form of the Rosuvastatin Adherence questionnaire (RAQ), Beliefs about Medicine Questionnaire - General (BMQ-G), and a Lifestyle questionnaire (LSQ) on disease understanding, lifestyle and treatment awareness. Patients in the Active group will also receive feedback on their daily rosuvastatin treatment as entered in the patient support tool.
* Control group: In this group the patients will have no additional support beyond the commonly practiced patient information, i.e. the patients will have no access to the smart phone-based patient support tool. However, a smart phone application will be used to prompt patients with the questions for the clinical evaluation (RAQ, BMQ-G and LSQ).

In this study, no rosuvastatin will be dispensed to the study participants i.e. patients will purchase their rosuvastatin prescription themselves as in normal practice. All assessments in this study (including blood sampling for the lipid profile) will not be used for guiding the treatment of patients in the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Female or male aged 18-80 years, diagnosed with dyslipidemia or hyperlipidemia at high risk and prescribed rosuvastatin

Dyslipidemia or hyperlipidemia defined as:

LDL-C≥2.6 mmol/L and TG<4.52mmol/L

High risk complies with any of the following:

* Documented cardiovascular disease (CVD) by invasive or non-invasive testing (such as coronary angiography, nuclear imaging, stress echocardiography, carotid plaque on ultrasound), previous myocardial infarction (MI), acute coronary syndrome (ACS), coronary revascularization [percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG)] and other arterial revascularization procedures, ischaemic stroke and peripheral arterial disease (PAD).
* Patients with type 2 diabetes, patients with type 1 diabetes with target organ damage (such as microalbuminuria).
* Patients with moderate to severe chronic kidney disease [(CKD), glomerular filtration rate (GFR) < 60 mL/min/1.73 m2].

  * Patients must have a smart phone that is compatible with the patient support tool and clinical evaluation questionnaire at their disposal and are comfortable with using of interactive smart phone applications. The required specification for the phone will be determined after completed testing.
  * Ability to read, understand and write Chinese.
  * Statin-naïve or with no statin use during the last 4 weeks prior to enrolment except in the event of patients may receive at most 7 doses of statins during current hospitalization before enrollment.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Previous enrolment or randomisation in the present study
* Participation in another clinical study with an investigational product or device during the last 30 days excluding prospective/retrospective register based studies that do not require any extra visits in addition to ordinary health care. Patients who withdraw from this study for any reason cannot re-enter the study.
* Patients in whom rosuvastatin is contraindicated i.e.

  * patients with hypersensitivity to rosuvastatin or any of the excipients.
  * patients with active liver disease including unexplained, persistent elevations of serum transaminases and have serum transaminase elevation exceeding 3 x the upper limit of normal (ULN).
  * patients with severe renal impairment (creatinine clearance <30 ml/min).
  * patients with myopathy.
  * patients receiving concomitant cyclosporin.
  * females during pregnancy and lactation and women of childbearing potential who are not using appropriate contraceptive measures.
* Significant medical or psychological condition that, in the opinion of the Investigator, would compromise the patient's safety or successful participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 885 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2016-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan C Carlsson, Study Director — AstraZeneca R&D
Locations (13):
- China (13):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Hangzhou
  - Research Site, Huzhou
  - Research Site, Nanchang
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Tianjin
  - Research Site, Waifang
  - Research Site, Wenzhou
  - Research Site, Wuhan

REFERENCES:
- [Background] Horne R, Weinman J. Patients' beliefs about prescribed medicines and their role in adherence to treatment in chronic physical illness. J Psychosom Res. 1999 Dec;47(6):555-67. doi: 10.1016/s0022-3999(99)00057-4. PMID 10661603

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 885 patients signed Inform Consent and were randomized in the study, 443 subjects in the active group and 442 subjects in the control group. 320 (72.2%) and 316 (71.5%) patients, respectively, completed the study. The overall completion rate was 71.9%. 31 patients (12 and 19 respectively) was not successful in receiving the relevant application.
Pre-assignment Details: A total of 885 patients were randomized (1:1) to two groups: an active group which received the smart phone-based patient support tool and a control application used for data collection only.
Groups:
- Active Group: receive the smart phone-based patient support tool
- Control Group: provided only the control application and not the smart phone-based patient support tool
Period: Overall Study
Arm/Group | Active Group | Control Group
Started | 443 | 442
Completed | 320 | 316
Not Completed | 123 | 126
Not completed — Severe non-compliance to protocol | 13 | 7
Not completed — Eligibility criteria not fullfilled | 7 | 3
Not completed — Withdrawal by Subject | 101 | 99
Not completed — Lost to Follow-up | 2 | 14
Not completed — Death | 0 | 3

BASELINE CHARACTERISTICS:
Population: The baseline characteristics were summarized based on the FAS, which comprised all randomized patients who received the study application successfully.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Group | Control Group | Total
Number analyzed (Participants) | 431 | 423 | 854
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (9.80) | 54.5 (9.51) | 54.6 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 154 | 315
  Male | 270 | 269 | 539
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 431 | 423 | 854
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 431 | 423 | 854
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Duration of Treatment
Description: The time from randomization to last patient reported visit (prior to the end-of-study visit) to a doctor to get a prescription for rosuvastatin plus the number of days of medicine provided in that last prescription.
Time Frame: limited to 169 days
Population: FAS
Measure: Mean (Standard Error); unit: days
Arm/Group | Active Group | Control Group
Number analyzed (Participants) | 431 | 423
days | 156.7 (2.24) | 146.0 (2.69)
Statistical Analysis 1: Comparison: Active Group vs Control Group; Test type: Superiority or Other; p = 0.0019, Log Rank

2. Secondary Outcome: Percentage of Fully Adherent Patients
Description: The number of patients who answered 'Yes' to Q4 of Rosuvastatin Adherence Questionnaire (RAQ) at all time points divided by the total number of randomized patients.
Time Frame: Up to 24 weeks
Population: FAS
Measure: Number; unit: % of patients
Arm/Group | Active Group | Control Group
Number analyzed (Participants) | 431 | 423
% of patients | 4.4 | 9.9
Statistical Analysis 1: Comparison: Active Group vs Control Group; Test type: Superiority or Other; p = 0.0017, Chi-squared

3. Secondary Outcome: Treatment Adherence
Description: The number of reported rosuvastatin tablets taken divided by the total number of days in the study.
Time Frame: Up to 24 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: % adherence
Arm/Group | Active Group | Control Group
Number analyzed (Participants) | 200 | 219
% adherence | 37.95 (32.916) | 58.19 (36.257)
Statistical Analysis 1: Comparison: Active Group vs Control Group; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -20.24, 95% CI 2-sided [-26.91 to -13.57], Standard Error of Mean 3.39

4. Post Hoc Outcome: Reported Treatment Adherence
Description: The number of reported rosuvastatin tablets taken divided by the total number of days reported during the treatment. This is eliminated any missing data from the calculation.
Time Frame: Up to 24 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: % adherence
Arm/Group | Active Group | Control Group
Number analyzed (Participants) | 200 | 219
% adherence | 94.63 (18.347) | 96.01 (14.316)
Statistical Analysis 1: Comparison: Active Group vs Control Group; Test type: Superiority or Other; p = 0.3939, t-test, 2 sided; Mean Difference (Final Values) = -1.38, 95% CI 2-sided [-4.56 to 1.80], Standard Error of Mean 1.60

5. Secondary Outcome: Percent Change in Low-Density Lipoprotein-Cholesterol (LDL-C) From Baseline
Description: Low-Density Lipoprotein-Cholesterol (LDL-C) change from baseline at the Week 24 assessment for subjects who completed 24 weeks of treatment
Time Frame: Baseline and Week 24
Population: FAS
Measure: Mean (Standard Error); unit: % change
Arm/Group | Active Group | Control Group
Number analyzed (Participants) | 303 | 303
% change | -21.09 (1.40) | -21.72 (1.40)
Statistical Analysis 1: Comparison: Active Group vs Control Group; Test type: Superiority or Other; p = 0.7514, ANCOVA; linear model including terms for randomized group and baseline LDL-C; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [-3.27 to 4.53], Standard Error of Mean 1.99

ADVERSE EVENTS:
Time Frame: 177±7 days
Description: This was an evaluation of the smart phone-based patient support tool, and rosuvastatin was not considered an investigational product for this study. There was no requirement to report AEs as part of the study, except the ones meeting the SAE criteria.
  Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Active Group | Control Group
Serious Adverse Events (participants affected / at risk) | 23/431 | 11/423
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Group (N=431) | Control Group (N=423)
Left carotid artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Right carotid artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (3) | 0 (0)
Cardiac insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac neurosis (Cardiac disorders) | 2 (2) | 0 (0)
Complete right bundle branch block (Cardiac disorders) | 1 (1) | 0 (0)
Coronary atherosclerosis (Cardiac disorders) | 0 (0) | 1 (1)
Coronary atherosclerotic heart disease (Cardiac disorders) | 4 (4) | 1 (1)
Coronary heart disease (Cardiac disorders) | 2 (2) | 5 (5)
Dilated cardiomyopathy (Cardiac disorders) | 1 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Persistent atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Unstable angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular premature beat (Cardiac disorders) | 1 (1) | 0 (0)
Macular edema (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 0 (0) | 1 (2)
Somatization disorder (General disorders) | 1 (1) | 0 (0)
Limb mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Acute renal insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The secondary endpoints Percentage of fully adherent patients and Treatment adherence may be impacted by the response frequency to the relevant questions. There is a tendency to a higher response frequency in the Control group in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No